CLINICAL TRIAL: NCT00443495
Title: First Into Man Administration of Chitin Microparticles: a Randomised,Double Blind,Placebo Controlled Parallel Group Upward Titration Evaluation of 3 Dose Levels Given Intr-Nasally Over 24 Hours,Followed by a Placebo Controlled,Randomised Parallel Group Evaluation of Safety and Biological Activity Over 7 Days in Subjects Suffering From Allergic Rhinitis
Brief Title: Phase I/IIa Study on Chitin Microparticles in Subjects Suffering From Allergic Rhinitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CMP Therapeutics Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMP/01/006; 06-505
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chitin microparticles by nasal route

SUMMARY:
Chitin microparticles (CMP) has been demonstrated in animal studies that have modelled allergic rhinitis to be effective against a wide range of common respiratory allergens. It is an immuneenhancer.

The primary purpose of the study is to demonstrate safety in a first into man study on 24 human volunteers. The secondary objective is to demonstrate efficacy by chosing subjects that demonstrate a response to a nasal allergen challenge using grass pollen.

The subjects are being given increasing doses of CMP, supplied as a nasal spray, for 7 days followed by a nasal allergen challenge with Timothy Grass Pollen extract. Over this period nasal symptom scores, eosinophil counts and cytokine measurements will be performed.

DETAILED DESCRIPTION:
Chitin microparticles are a special preparation of chitin. This a long chain polysaccaride derived from shells of the North Atlantic shrimp. CMP acts a an immunenhancer which improve immune function by stimulating macrophages and other cells such as T-helper lymphocytes, (Th cells). In allergies there is an imbalance between Th1 and Th2 cells. Imuneenhancers shift the balance in favour of Th1 cells. The immunomodulatory properties of CMP have been demonstrated in animal models against a wide range of respiratory allergens. There have been no indications of toxic side effects in animal models.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 50 years of age inclusive with a history of symptoms of allergic rhinitis within the previous two years.
2. Subjects must be free from clinically significant cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
3. Forced expiratory volume over one second (FEV1) within normal limits (≥ 90% of predicted, ECCS 1993).
4. Asymptomatic at screening as characterized by:

   1. Normal appearing nasal mucosa with no active allergic rhinitis.
   2. A pre-nasal allergen challenge total nasal symptom score sheet on study entry so that subjects produce a score of <2 at screening.
5. Non smokers for at least the past 12 months with a pack history ≤ 1 pack years (Pack years = (n of cigarettes smoked/day/20) x n of years smoked).
6. An increase in nasal symptom score of between 4 and 10 following screening nasal allergen challenge.
7. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
8. Available to complete the study.
9. Negative urinary drugs of abuse screen, determined at screening and in the 24 hours before the first dose of study medication.
10. Negative carbon monoxide test (smokerlyzer) determined at screening and in the 24 hours before the first dose of study medication.
11. Clinically normal vital signs and 12-lead electrocardiogram (ECG), determined at screening.
12. A body mass index (Quetlet index) in the range of 18.00 to 30.9.

Exclusion Criteria:

1. Perennial rhinitis.
2. Upper respiratory tract infection within 2 weeks of the first dose of study medication.
3. Medical conditions likely to affect the outcome of the study in the opinion of the investigator.
4. Nasal conditions likely to affect the outcome of the study in the opinion of the investigator, i.e. nasal septal perforations, nasal polyps, sinus disease, chronic nasal obstruction, or other nasal diseases.
5. Presence of any respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function (defined as ≥ 90% predicted for height and age, ECCS 1993).
6. History of immunotherapy in the past 3 years or currently on an immunotherapy treatment course including inhaled or local corticosteroids in the past 28 days.
7. Any infirmity, disability, or geographic location which, in the opinion of the principal investigator, would limit compliance with the protocol.
8. Infection of the upper airways/lower airways, sinus, or ear, including viral infections in the 14 days prior to screening and at the start of the treatment period.
9. Clinically significant abnormality in clinical laboratory tests at screening as determined by the principal investigator.
10. Inability to tolerate lavage correctly with a preliminary nasal lavage at screening.
11. Participation in a study with a new molecular entity during the previous four months or any other trial during the previous three months.
12. The subject regularly, or on average, drinks more than four units of alcohol per day.
13. Testing positive for hepatitis C antibody or hepatitis B surface antigen or for HIV.
14. Receipt of prescribed or over the counter medication (including herbal remedies and dietary supplements) within 14 days of the first dose of test article and for the duration of the trial (with the exception of paracetamol up to 2g daily). In particular, all antihistamines, chromoglycate and steroids are prohibited during this period.
15. Inability to communicate well with the investigator (i.e., language problem, poor mental development or impaired cerebral function).
16. Donation of 450 mL or more blood within the previous 12 weeks.
17. A history of hypersensitivity and/or idiosyncrasy to any of the test compounds or excipients employed in this study.
18. Subjects with clinical features suspicious of tuberculosis - weight loss, pyrexia, haemoptysis, purulent sputum, previous abnormal chest X-ray will be excluded from the study.
19. Clinical evidence of autoimmune disease.
20. Allergy to seafood.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-10; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Warrington, MA MD FRCP FFPM, Principal Investigator — Hammersmith Medicines Research